CLINICAL TRIAL: NCT00969124
Title: Impact of Experience With the Third Eye Retroscope on Detection Rates and Withdrawal Times During Colonoscopy
Brief Title: Impact of Experience on Results With the Third Eye Retroscope
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Avantis Medical Systems (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Avantis TER 08-07
Record Dates: First submitted 2009-08-27; First posted 2009-09-01 (Estimated); Results first posted 2017-07-26 (Actual); Last update posted 2017-07-26 (Actual); Status verified 2017-06

CONDITIONS: Colorectal Neoplasms
Keywords: colonoscopy; polyps; adenomas; miss rates
MeSH Terms: conditions — Colorectal Neoplasms; Polyps; Adenoma

STUDY DESIGN:
Masking Description: Open Label
Oversight: Data Monitoring Committee: No

ARMS (1):
- Third Eye Retroscope (Experimental): All subjects underwent the same intervention, consisting of examination of the colon using a colonoscope along with the Third Eye Retroscope device, with removal of any polyps that were detected during the procedure.
  Interventions: Device: Third Eye Retroscope

INTERVENTIONS:
Device: Third Eye Retroscope — Third Eye Retroscope is used in conjunction with a standard colonoscope while performing colonoscopy

SUMMARY:
The Third Eye Retroscope is a device that can be used with a colonoscope to improve the ability of a physician to see areas of the colon that may be hidden from the view of the colonoscope.

Previous studies have shown that physicians are able to detect additional polyps when they use the device along with the colonoscope. The purpose of this study is to determine whether physicians can detect greater numbers of additional polyps as they gain in experience with the device.

DETAILED DESCRIPTION:
Purpose: This study is intended to determine characteristics of the "learning curve" for use of the Third Eye Retroscope during colonoscopy, both in terms of efficacy for detection of abnormalities in the colon and time-efficiency for endoscopists

Device Description: The Third Eye Retroscope is an auxiliary imaging device that is designed to allow visualization of "hidden areas" during colonoscopy by providing an additional, retrograde view that complements the forward view of the colonoscope.

After a standard colonoscope has been advanced to the cecum, the Third Eye Retroscope is inserted through the instrument channel of the colonoscope. As it emerges from the distal tip of the colonoscope, the Third Eye Retroscope automatically bends 180 degrees to form a "J" shape. Its sensor then provides a continuous retrograde view of the colon throughout the process of withdrawal of the colonoscope.

The retrograde view assists the endoscopist in visualizing the proximal aspect of haustral folds and rectal valves, as well as the areas behind flexures and the ileocecal valve. With this additional point-of-view, the endoscopist may be able to detect lesions that can be missed by the forward-viewing colonoscope.

Study Design: Patients who are scheduled for colonoscopy will be recruited to the study and examined with the Third Eye Retroscope in conjunction with a standard colonoscope. For each polyp that is found, the endoscopist will indicate whether it could be seen with the colonoscope, or if it could be found with the colonoscope only because it was first detected with the Third Eye.

Each investigator will perform colonoscopies on 20 patients, who will be segmented into four quartiles according to the order of their procedures. Mean results for the quartiles will be compared in order to evaluate the learning curve for Third Eye colonoscopy.

ELIGIBILITY:
Inclusion Criteria:

1. The patient is undergoing colonoscopy for screening, for surveillance in follow-up of previous polypectomy or for diagnostic workup;
2. The patient must understand and provide written consent for the procedure.

Exclusion Criteria:

1. Patients with a history of colonic resection;
2. Patients with inflammatory bowel disease;
3. Patients with a personal history of polyposis syndrome;
4. Patients with suspected chronic stricture potentially precluding complete colonoscopy;
5. Patients with diverticulitis or toxic megacolon;
6. Patients with a history of radiation therapy to abdomen or pelvis.
7. Patients who are currently enrolled in another clinical investigation in which the intervention might compromise the safety of the patient's participation in this study.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 328 (Actual)
Dates: Start 2009-01; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel C DeMarco, MD, Principal Investigator — Baylor Health Care System
Locations (9):
- United States (9):
  - Florida Hospital, Celebration, Florida
  - University of Chicago, Chicago, Illinois
  - NorthShore University HealthSystem, Evanston, Illinois
  - University of Massachusetts, Worcester, Massachusetts
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Parkland Hospital, Dallas, Texas
  - Baylor University Medical Center, Dallas, Texas
  - S.W. Fort Worth Endoscopy Center, Fort Worth, Texas
  - North Hills Hospital, North Richland Hills, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] DeMarco DC, Odstrcil E, Lara LF, Bass D, Herdman C, Kinney T, Gupta K, Wolf L, Dewar T, Deas TM, Mehta MK, Anwer MB, Pellish R, Hamilton JK, Polter D, Reddy KG, Hanan I. Impact of experience with a retrograde-viewing device on adenoma detection rates and withdrawal times during colonoscopy: the Third Eye Retroscope study group. Gastrointest Endosc. 2010 Mar;71(3):542-50. doi: 10.1016/j.gie.2009.12.021. PMID 20189513

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Third Eye Retroscope
Started | 328
Completed | 298
Not Completed | 30
Not completed — Protocol Violation | 2
Not completed — Inadequate bowel preparation | 15
Not completed — Inability to reach cecum | 9
Not completed — Previously unrecognized disease | 3
Not completed — Technical error | 1

BASELINE CHARACTERISTICS:
Population: Per-protocol population of patients for whom the colonoscopy procedure was completed using the Third Eye Retroscope, not including the 30 who were withdrawn due to reasons stated above.
Arm/Group | Third Eye Retroscope
Number analyzed (Participants) | 298
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.8 (11.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 154
  Male | 144
Region of Enrollment [Number; unit: participants]
  United States | 298
Indication for colonoscopy procedure (screening, surveillance or diagnostic) [Number; unit: participants]
  Screening | 164
  Surveillance | 62
  Diagnostic | 72

OUTCOME MEASURES:

1. Primary Outcome: Detection Rates for Adenomas
Description: Adenomas detected with the colonoscope alone vs. with the Retroscope
Time Frame: During the colonoscopy procedure (up to 1 hour, average 25 minutes)
Measure: Number; unit: Adenomas
Arm/Group | Third Eye Retroscope
Number analyzed (Participants) | 298
Adenomas
  Adenomas detected with colonoscope alone | 100
  Additional adenomas detected with Retroscope | 16

2. Primary Outcome: Detection Rates for All Polyps
Description: All polyps detected with the colonoscope alone vs. with the Retroscope
Time Frame: During the colonoscopy procedure (up to 1 hour, average 25 minutes)
Measure: Number; unit: All polyps
Arm/Group | Third Eye Retroscope
Number analyzed (Participants) | 298
All polyps
  All polyps detected with colonoscope alone | 182
  Additional all polyps detected with Retroscope | 27

3. Secondary Outcome: Time Spent During Withdrawal Phase and Total Procedure
Description: Time in minutes for withdrawal phase of procedure and for total procedure
Time Frame: During the colonoscopy procedure (up to 1 hour, average 25 minutes)
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Third Eye Retroscope
Number analyzed (Participants) | 298
minutes
  Average withdrawal time | 9.9 (4.1)
  Average total procedure time | 24.7 (9.7)

ADVERSE EVENTS:
Time Frame: 48-hour telephone follow-up to assess for post-procedural complications
Arm/Group | Third Eye Retroscope
Serious Adverse Events (participants affected / at risk) | 0/298
Other Adverse Events (participants affected / at risk) | 0/298

LIMITATIONS AND CAVEATS:
No randomization or blinding and no separate control group. Determinations regarding adequacy of bowel cleansing and whether each polyp could have been detected with the colonoscope alone involved a judgement by the endoscopist.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No